CLINICAL TRIAL: NCT01447875
Title: The Effects of Propofol and Dexmedetomidine Infusion on the Fluid Responsiveness in Critically Ill Patients
Brief Title: The Effects of Sedative on the Fluid Responsiveness in Critically Ill Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Tao Yu, clinical doctor, Southeast University, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2011ZDLLKY02.1
Record Dates: First submitted 2011-10-05; First posted 2011-10-06 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2012-05

CONDITIONS: Shock; Sepsis
MeSH Terms: conditions — Shock; Sepsis | interventions — Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Passive Leg Raising — elevation of both legs to a 45 degrees for about 1-2 minute before sedation
  Other Names: Passive Leg Raising testing
Drug: propofol or mexmedetomidine

SUMMARY:
Hypotension and bradycardia are often observed following induction of dexmedetomidine or propofol sedation.Cardiac preload decrease by sedative agents was often considered as one of main causes for this hypotension.The investigators hypothesized that hypotension after induction of sedation is caused by decrease of preload by sedative agents,and passive leg raising (PLR)test could predict this event.Dexmedetomidine or propofol infusion in patients with circulatory failure decrease cardiac preload and enhance preload-dependency and fluid responsiveness.

DETAILED DESCRIPTION:
In this clinical trial,the investigators hypothesized dexmedetomidine or propofol infusion in patients with circulatory failure decrease cardiac preload and enhanced preload-dependency and fluid responsiveness,and PLR induced pulse pressure variation (PLR-ΔPP) could predict the hypotension during dexmedetomidine induction in critically ill patients.Before dexmedetomidine or propofol infusion, the investigators will conduct passive leg raising test. At first, the patient's trunk was elevated 45 degrees for the first set of measurements. Then, the lower limbs were raised to a 45° angle while the patient's trunk was lowered to a supine position to measure peak BP (usually within 30-90 s). Hemodynamic profiles planned to be measured are SBP, DBP, CVP and HR.Sedation was induced with a dexmedetomidine 0.5μg/kg over 10 min loading, followed by a maintenance infusion of 0.2-0.7 μg/kg/h for one hour. The dose of propofol was titrated targeting the Richmond agitation sedation scale (RASS) ranged from -2 to -1 (bispectral index: 60-75).Hypotension was defined as a SBP less than 80 mmHg or DBP was less than 50 mmHg, or greater than 30% decrease from baseline for longer than 60 s. Bradycardia was defined a HR 50 /min or greater than 30% change from baseline for longer than 60 s. Receiver operator characteristic curve analysis was performed to evaluate sensitivity and specificity of the value PLR-ΔPP to detect patients at high risk of hypotension.

ELIGIBILITY:
Inclusion Criteria:

* patients with at least one of the clinical manifestations of acute circulatory failure; patients undergoing dexmedetomidine or propofol infusion

Exclusion Criteria:

* deep venous thrombosis or elastic compression stocking
* an increase in the intra-abdominal pressure confirmed by clinical examination
* serious central nervous system pathology (head trauma, severe dementia, acute stroke, uncontrolled seizures)
* severe liver disease(Child-Pugh class C)
* unstable angina or acute myocardial infarction
* left ventricular ejection fraction less than 30%
* heart rate(HR) less than 50/min, heart block with second- or third degree
* systolic blood pressure (SBP) less than 90 mmHg despite 2 vasopressors infusion continuously before the begin of dexmedetomidine infusion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
the area under ROC curve to predict hypotension | 60 min around passive leg raising test
  area under ROC curve of blood pressure changes during PLR to predict hypotension during sedation

CONTACTS AND LOCATIONS:
Overall Officials: Tao Yu, Study Director — Nanjing Zhong-Da Hospital, Southeast University
Locations (1):
- Nanjing Zhong-Da Hospital, Southeast University School of Medicine, Nanjing, China